CLINICAL TRIAL: NCT05665010
Title: Precise Stratification of Genetic Risk of Ovarian Function Impairment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Shixuan Wang, Professsor, Tongji Hospital
Other Study IDs: TJ-IRB20211016-SOA
Record Dates: First submitted 2022-11-30; First posted 2022-12-27 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Premature Ovarian Insufficiency; Diminished Ovarian Reserve; Early Menopause
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- premature ovarian insufficiency: Patients with premature ovarian insufficiency (female age <40 years, menopause or menstrual rarity for 4 months, basal FSH > 25 IU / L for two consecutive intervals of more than 4 weeks)
  Interventions: Other: Genetic susceptibility
- declined ovarian function: Patients with diminished ovarian reserve(women before 40 years old; the number of antral follicles in both ovaries is less than 6, AMH < 1.1ng/ml, and basal FSH > 10 IU / L, which meets one of the three requirements)；Female with menopause between the age of 40 and 45.
  Interventions: Other: Genetic susceptibility

INTERVENTIONS:
Other: Genetic susceptibility — Genetic susceptibility increases the risk of ovarian injury

SUMMARY:
Aging is a common problem in human society at present. The fertility decline, perimenopausal symptoms and senile diseases caused by ovarian aging seriously affect women's own health, offspring's health, family and social stability, and endanger national population security. Accurate stratification of genetic risk of ovarian aging has practical significance. Early and accurate identification of high-risk groups of premature ovarian aging can help such women to start early protection of ovarian function, preserve fertility to a greater extent, improve fertility quality, and also be conducive to early prevention and treatment of other systemic diseases and prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Women who meet the diagnosis of premature ovarian insufficiency (POI), diminished ovarian reserve (DOR) or early menopause and hope to find out the risk of premature ovarian impairment and clarify the cause of premature ovarian impairment;

   1. premature ovarian insufficiency (POI): the age of female is less than 40 years old, with menopause or sparse menstruation for 4 months, and basal FSH > 25IU / L for two consecutive times with an interval of more than 4 weeks.
   2. Diminshed ovarian reserve (DOR): before the age of 40, the number of antral follicles in both ovaries is less than 6, or AMH is less than 1.1ng/ml, or basal FSH is greater than 10 IU/L.
   3. Early menopause: women who enter menopause between the age of 40 and 45.
2. Informed consent, voluntary test.

Exclusion Criteria:

1. Chromosome karyotype abnormality;
2. Iatrogenic ovarian injury: history of radiotherapy, chemotherapy (reproductive toxic drugs such as alkylating agents) and ovarian surgery;
3. Ovarian mass: there is abnormal echo in the ovary under ultrasound, and the maximum diameter is greater than 4cm.
4. Pregnant and lactating women;
5. Polycystic ovary syndrome, hyperprolactinemia, hyperandrogenemia, hypothyroidism, adrenal dysfunction and other endocrine diseases affect ovulation;
6. Patients with cardiovascular, liver, kidney, hematopoietic system and other serious primary diseases and psychosis;
7. Patients who are participating in other clinical trials or have participated in other clinical trials in the past month;
8. Other patients determined by the investigator to be unsuitable for participation in this study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: A multi regional ovarian aging cohort of Chinese population, including 500 patients with premature ovarian insufficiency, 500 patients with diminished ovarian reserve or early menopause.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Genetic variants | 2 year
  Genetic variants that differed significantly between participants and the general population

SECONDARY OUTCOMES:
Menopause age | One year after the last menstruation
  Menopause for more than one year

CONTACTS AND LOCATIONS:
Overall Officials: Shixuan Wang, Doctor, Study Chair — Tongji Hospital, Affiliated to Tongji Medical College of Huazhong University of Science and Technology
Locations (18):
- China (18):
  - Fujian maternal and Child Health Hospital, Fuzhou, Fujian
  - Guangdong maternal and Child Health Hospital, Guangzhou, Guangdong
  - Guangdong Provincial People's Hospital, Guanzhou, Guangdong
  - Shijiazhuang maternity hospital, Shijiazhuang, Hebei
  - The Third Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of science and technology, Wuhan, Hubei
  - Central South Hospital of Wuhan University, Wuhan, Hubei
  - Hubei maternal and Child Health Hospital, Wuhan, Hubei
  - Liyuan Hospital Affiliated to Tongji Medical College of Huazhong University of science and technology, Wuhan, Hubei
  - People's Hospital of Wuhan University, Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - Changsha maternal and Child Health Hospital, Changsha, Hunan
  - The First Affiliated Hospital of Suzhou University, Suzhou, Jiangsu
  - Jiangxi maternal and Child Health Hospital, Nanchang, Jiangxi
  - Northwest women and children's Hospital, Xi’an, Shanxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Affiliated Hospital of Yunnan University, Kunming, Yunnan
  - Hospital of Obstetrics and Gynecology affiliated to Medical College of Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ma W, Ye S, Tian L, Liu M, Wang R, Yang X, Wang M, Fu F, Ren W, Dang L, Wang T, Wang W, Wang S, Sun Y, Li Y. Association of LHCGR rs2293275 genotype with ovarian aging in Chinese women: a multicenter population-based study. Reprod Biol Endocrinol. 2025 Mar 15;23(1):41. doi: 10.1186/s12958-025-01375-2. PMID 40089715